CLINICAL TRIAL: NCT04137081
Title: Managing Risk at Its Source: Reducing Clinician Burnout Through Digital Therapeutic Delivery of Mindfulness Training
Brief Title: Unwinding Physician Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Judson Brewer, Principal Investigator, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H00014985
Record Dates: First submitted 2019-10-22; First posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Anxiety; Burnout, Professional
Keywords: Physicians
MeSH Terms: conditions — Anxiety Disorders; Burnout, Professional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- App-based mindfulness training (Experimental): The Unwinding Anxiety program is delivered via a smartphone-based platform, which includes a progression through 30+ daily modules of brief didactic and experience-based mindfulness training (videos and animations), app-triggered check-ins to encourage engagement, and user-initiated guided mindfulness exercises to help disrupt worry cycles in the moment.
  Interventions: Behavioral: App-based mindfulness training

INTERVENTIONS:
Behavioral: App-based mindfulness training — Unwinding Anxiety is an app-based mindfulness training program which includes a progression through 30+ daily modules. Each module's training is delivered via short video tutorials and animations (~10 min/day). Each training builds on the previous one; modules are 'locked' so that they can only be viewed at a pace of 1/day (previous modules can be reviewed at any time). A built-in self-assessment is taken after every seven modules to ensure key concepts are learned before moving on with automated suggestions on which modules to repeat based on self-assessment results. User-initiated guided practices range from short exercises (30 seconds) to manage anxiety the moment it arises to formal guided meditations (up to 15 minutes), and can be accessed at any time.

SUMMARY:
The purpose of this study is to test an app-based mindfulness training program to see if it can reduce anxiety and burnout in physicians.

DETAILED DESCRIPTION:
In this study, 50 clinicians will be provided access to the Unwinding Anxiety program. The intervention period will last 3 months and changes in anxiety and burnout along with program engagement will be assessed at baseline, 1 month, and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Currently employed as a physician
* Direct patient interaction
* Owns a smartphone
* Endorsed anxiety based on answering yes to following questions:

  1. Do you feel nervous, anxious, or on edge?
  2. Do you feel you worry too much about different things?
* Endorsed willingness to use smartphone app for 10+ minutes/day for 30 days
* Endorsed willingness to complete online surveys

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Changes in anxiety | 1 month
  Generalized Anxiety Disorder 7-item (GAD-7) questionnaire will be used to assess anxiety. The GAD-7 uses a 4-point Likert scale where 0 is "Not at all" to 3 "Nearly every day". Scores can range from 0 to 21 and higher scores indicate increasing severity of anxiety.

SECONDARY OUTCOMES:
Changes in burnout | 1 month
  Two, single-item questions from the emotional exhaustion and cynicism domains of the Maslach Burnout Inventory will be used to assess burnout. Both questions are on a 7-point Likert scale where 0 is "never" and 7 is "every day". Scores can range from 0 to 7 for each domain and higher scores indicate increasing levels of burnout.
Program engagement | 1 month
  Program engagement will be assessed based on the number of modules completed. The program has 30 modules therefore scores scan range from 0 to 30 modules.

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — UMass Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roy A, Druker S, Hoge EA, Brewer JA. Physician Anxiety and Burnout: Symptom Correlates and a Prospective Pilot Study of App-Delivered Mindfulness Training. JMIR Mhealth Uhealth. 2020 Apr 1;8(4):e15608. doi: 10.2196/15608. PMID 32234708